CLINICAL TRIAL: NCT01274273
Title: A Randomized Phase II Trial of IL-2/IFN-α Plus Bevacizumab Versus IL-2/IFN-α in Metastatic Renal Cell Carcinoma (mRCC) - Danish Renal Cancer Group (DARENCA) Study-1
Brief Title: Study of Interleukin-2, Interferon-alpha and Bevacizumab in Metastatic Kidney Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Danish Renal Cancer Study Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DARENCA-1
Record Dates: First submitted 2010-06-29; First posted 2011-01-11 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2012-08

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Bevacizumab; interleukin-2; interferon-alpha
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Interleukin-2; aldesleukin; Interferon alpha-2; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interleukin-2, interferon, bevacizumab (Experimental)
  Interventions: Drug: Bevacizumab
- Interleukin-2 and interferon-alfa (Active Comparator)
  Interventions: Drug: Interleukin-2; Drug: Interferon Alfa-2b

INTERVENTIONS:
Drug: Interleukin-2 — 2.4 MIU/m2 s.c. two times daily, 5 days per week, weeks 1 and 2, every 28-day-cycle, for a maximum of 9 cycles (i.e.for a maximum of 9 months).
  Other Names: Aldesleukin
  Arms: Interleukin-2 and interferon-alfa
Drug: Interferon Alfa-2b — IFN-alfa given as one priming-week of daily IFN 3.0 MIU, followed by up to 9 treatment cycles (i.e. for a maximum of 9 months) with IFN-alfa 3.0 MIU as a fixed dose s.c. once daily - 5 days per week.
  Other Names: IntronA
  Arms: Interleukin-2 and interferon-alfa
Drug: Bevacizumab — Bevacizumab doses of 10 mg per kilogram of body weight, given every two weeks i.v. until disease progression, unacceptable toxicity, withdrawal of consent or a maximum of 1 year following obtaining no evidence of disease (NED).
  Other Names: Avastin
  Arms: Interleukin-2, interferon, bevacizumab

SUMMARY:
The purpose of this study is to determine whether interleukin-2, interferon-alpha in combination with bevacizumab are effective in the treatment of metastatic renal cell carcinoma (mRCC).

DETAILED DESCRIPTION:
Bevacizumab as monotherapy has effect in metastatic renal cell carcinoma (mRCC). Bevacizumab in combination with interferon-alfa (IFN-α) has significant efficacy in mRCC and has been approved by EMA and FDA.

The present study will assess whether the combination of Interleukin-2 (IL-2) and IFN-α with bevacizumab may add efficacy in patients with mRCC with a tolerable safety profile.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Patient must be willing and able to comply with the protocol.
3. Age ≥ 18 years.
4. Histologic og cytologic biopsy proven locally advanced or metastatic renal cell carcinoma, considered non-candidates for curative surgery. Nephrectomy is not mandatory.
5. Patient with renal cell carcinoma (RCC) with a clear-cell histologic component confirmed by local pathology review.
6. Females with a negative serum pregnancy test unless childbearing potential can be otherwise excluded
7. Fertile women of childbearing potential (<2 years after last menstruation) and men must use effective means of contraception
8. Memorial-Sloan-Kettering-Cancer-Centre favourable- and intermediate prognostic group.
9. Measurable or non-measurable disease (as per RECIST1.1 criteria)
10. Karnofsky Performance status of 70% or higher.
11. Life expectancy greater than 4 months.
12. The required laboratory values at baseline are as follows:

Haematology:

WCC ≥ 3.0 x 109/L, Platelet count ≥ 100 x 109/L, Haemoglobin ≥ 6.2 mmol/l, (INR) ≤ 1.5, APTT ≤ 1.5 x ULN

Biochemistry:

Total bilirubin ≤ 1.5 x upper limit of normal (ULN), AST, ALT ≤ 2.5 x ULN in patients without liver metastases, ≤ 5 x ULN in patients with liver metastases, Serum Creatinine ≤ 150 micromol/L

-

Exclusion Criteria:

1. Prior systemic treatment for metastatic RCC disease
2. Major surgical procedure, open surgical biopsy, or significant traumatic injury within 28 days prior to randomization.
3. Serious non-healing wound, ulcer or bone fracture.
4. Evidence of current central nervous system (CNS) metastases or spinal cord compression. Patient must undergo an MRI or CT scan of the brain (with contrast, if possible) within 28 days prior to randomization.
5. Seizure(s) not controlled with standard medical therapy.
6. Dipstick urine test of protein ≥ 2+.
7. Other malignancies within 5 years prior to randomization (other than curatively treated basal cell carcinoma of the skin and/or in situ carcinoma of the cervix).
8. Evidence of bleeding diathesis or coagulopathy.
9. Ongoing or recent (within 10 days prior to study treatment start) need for full therapeutic dose of oral anticoagulants or chronic daily treatment with aspirin. Low molecular weight heparin are allowed
10. Uncontrolled hypertension (≥ 160 mm Hg systolic and/or ≥ 100 mm Hg diastolic) while receiving chronic medication.
11. Clinically significant (i.e. active) cardiovascular disease, for example cerebrovascular accidents (≤ 6 months before randomisation), myocardial infarction (≤ 6 months before randomisation), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication.
12. Recent (within the 30 days prior to randomization) treatment with another investigational drug or participation in another investigational study.
13. Chronic treatment with corticosteroids (dose of ≥ 10 mg/day methylprednisolone equivalent), excluding inhaled steroids.
14. History or presence of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or patient at high risk from treatment complications.
15. Known hypersensitivity to interleukin-2, Interferon, alfa or bevacizumab.

Serial blood test, serial tumor biopsies and serial dynamic contrast-enhanced imaging will be obtained as part of a translational research program integrated in the clinical trial.

Part(s) of the translational research program may be omitted in the individual patient due to practical, technical or safety reasons, without having consequences for participating in the additional translational research investigations or the clinical part of the study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2009-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival, PFS | This is defined as the time between date of randomisation and the first date of documented disease progression or date of death due to any cause.

SECONDARY OUTCOMES:
Response rate, RR | Overall response rate as assessed by the RECIST 1.1 criteria. An overall response is defined as a confirmed complete response (CR) or confirmed partial response (PR).
Overall survival, (OS) | Overall survival is defined as the time between date of randomisation and the date of death due to any cause.
Duration of response | Duration of response is defined as the time between the date a response (CR or PR) was first seen until date of progression.
Time to progression, (TTP) | Time to progression is defined as time between date of randomisation and date of documented progression.
Time to treatment failure, (TTTF) | see below
  Time to treatment failure is defined as time between date of randomisation and date of insufficient therapeutic response (including disease progression), death, withdrawal of treatment due to adverse events or laboratory abnormality, or withdrawn informed consent.
Tolerability | see below
  Toxicity is recorded according to CTCAE v3.0
Frequency of surgical resection of residual disease | see below
  This is calculated as number of patients having surgical resection of residual disease compared with the total number of treated patients.
Frequency of no evidence of disease (NED) | see below
  This is calculated as the total number of patients having no evidence of disease as a result of CR to treatment, or as a result of PR/SD to treatment followed by surgical resection of residual disease, compared with the total number of treated patients.
To explore the immunomodulatory effect of therapy in serial blood samples and serial tumor core biopsies and to correlate these biomarkers with outcome | see below
  Blood tests and core biopsies from accessible tumor lesions will be obtained at baseline, after cycle 1 and at PD.
  Blood analyses will include assessment of dendritic cells, FoxP3+ regulatory T-cells, NK-cells, T-subsets, neutrophils, monocytes, cytotoxic activity and antibody-dependent cellular cytotoxicity (ADCC).
  Tumor analyses will include assessment of intratumoral immune cells, markers related to HIF accumulation and CD34+ microvessel density.
To assess dynamic contrast-enhanced imaging as a potential biomarker. | see below
  Dynamic contrast-enhanced imaging (CT, MRI, and US) will be obtained at baseline, week 5 and at routine tumor assessments, if appropriate, for estimation of tumor blood perfusion change.
  An exploratory analysis to identify any potential relationship between each of these assessments and outcome (progression free survival, survival, time to progression, response rate and safety) will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Frede Donskov, MD, DMSc, Principal Investigator — Aarhus University Hospital; Poul Geertsen, MD, PhD, Study Chair — University of Copenhagen
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus, Aarhus
  - Herlev University Hospital, Herlev, Herlev

REFERENCES:
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] Drljevic-Nielsen A, Rasmussen F, Nielsen PS, Stilling C, Thorup K, Mains JR, Madsen HHT, Donskov F. Prognostic value of DCE-CT-derived blood volume and flow compared to core biopsy microvessel density in patients with metastatic renal cell carcinoma. Eur Radiol Exp. 2021 Jul 30;5(1):32. doi: 10.1186/s41747-021-00232-2. PMID 34327591
- [Derived] Donskov F, Jensen NV, Smidt-Hansen T, Brondum L, Geertsen P. A randomized phase II trial of interleukin-2 and interferon-alpha plus bevacizumab versus interleukin-2 and interferon-alpha in metastatic renal-cell carcinoma (mRCC): results from the Danish Renal Cancer Group (DaRenCa) study-1. Acta Oncol. 2018 May;57(5):589-594. doi: 10.1080/0284186X.2018.1433324. Epub 2018 Feb 2. PMID 29392960